CLINICAL TRIAL: NCT03319368
Title: Implementation of a Novel Strategy to Prevent Staphylococcus Aureus (SA) Acquisition in Community-Based Nursing Homes to Prevent Invasive SA Infection - Feasibility and Pilot to Guide a Multicenter Stepped Wedge Cluster Trial
Brief Title: Preventing the Spread of Infection in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mary-Claire Roghmann, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00077879
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Targeted gown and glove use (Experimental): Additional gowns and gloves used for high risk care activities
  Interventions: Other: Targeted gown and glove use

INTERVENTIONS:
Other: Targeted gown and glove use — Gown and glove use for high risk care activities in high risk residents

SUMMARY:
This study evaluates the feasibility of targeting more frequent gown and glove use for specific high risk moments of care in specific nursing home residents in order to prevent Staphylococcus aureus (SA) acquisition and infection.

DETAILED DESCRIPTION:
Nursing homes are settings with a high rate of Staphylococcus aureus (SA) acquisition, which leads to infection, particularly for short stay residents. The current standard of care for preventing SA acquisition and SA infection in nursing homes is Standard Precautions (gowns and gloves for anticipated contact with blood, body fluids, skin breakdown or mucous membranes) for all residents.

The investigators propose a feasibility study of a novel strategy, the addition of targeted gown and glove use, to prevent SA acquisition and SA infection in residents of nursing homes. Rather than wearing gowns and gloves for all care activities to prevent transmission, gown and glove use can be targeted to specific high risk "moments" of care for specific high risk residents. High risk "moments" for gown and glove use are care activities most likely to transmit SA based on prior research. Residents with chronic wounds and medical devices are: 1) most likely to be colonized with SA; 2) most likely to acquire SA; 3) most likely to transmit SA to healthcare worker clothing and hands; and 4) most likely to develop a SA infection based on prior research and thus would be considered high risk residents.

The investigators will perform a quasi-experimental (before-after) study of this intervention, targeted gown and glove use, at two community-based nursing homes to demonstrate its feasibility and evaluate its effect on SA acquisition and SA infection rates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Reside in a participating nursing home

Exclusion Criteria:

* Identified by nursing home staff as combative or with other behavioral problems which could lead to agitation if approached by project staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lorien Riverside, Belcamp, Maryland
  - Lorien Mays Chapel, Lutherville-Timonium, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lydecker AD, Osei PA, Pineles L, Johnson JK, Meisel J, Stine OC, Magder L, Gurses AP, Hebden J, Oruc C, Mody L, Jacobs Slifka K, Stone ND, Roghmann MC. Targeted gown and glove use to prevent Staphylococcus aureus acquisition in community-based nursing homes: A pilot study. Infect Control Hosp Epidemiol. 2021 Apr;42(4):448-454. doi: 10.1017/ice.2020.1219. Epub 2020 Oct 20. PMID 33077004

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Long stay residents (n=42) were enrolled in the study specifically to examine if they transmitted S. aureus to short stay residents for the secondary outcome measure. They were excluded from all other study analyses.
Groups:
- Baseline Period: Normal, day-to-day usage of gowns and gloves by health care workers in nursing homes.
- Intervention Period: Targeted gown and glove use by health care workers in the nursing home. Gowns and gloves were worn when providing high risk care to high risk residents.
Period: Overall Study
Arm/Group | Baseline Period | Intervention Period
Started | 158 | 167
Completed | 101 | 121
Not Completed | 57 | 46
Not completed — Discharge swabs not collected from resident | 57 | 46

BASELINE CHARACTERISTICS:
Population: Participants who had both admission and discharge swabs collected during the study period. Both sets of swabs need to be collected to assess for acquisition of Staph aureus.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Period | Intervention Period | Total
Number analyzed (Participants) | 101 | 121 | 222
Age, Customized [Count of Participants; unit: Participants] — Age was not collected for this study.
  Participants | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/Gender was not collected for this study.
  Participants | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Co-colonized with MRSA and MSSA on admission swabs [Count of Participants; unit: Participants] — Participants who are colonized with both MRSA (methicillin resistant Staphylococcus aureus) and MSSA (methicillin susceptible Staphylococcus aureus) on their admission swabs. Swabs were collected from the anterior nares and inguinal fold.
  Participants | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rates of Staphylococcus Aureus Acquisition: Percentage of Short Stay Participants Who Acquired MRSA or MSSA (or Both) During the Study Period
Description: Rates of Staphylococcus aureus acquisition in the baseline and intervention periods: Participants were swabbed in the anterior nares and inguinal fold at nursing home admission (or start of study period) and again at discharge (or end of study period). This is the percentage of participants who acquired MRSA or MSSA (or both) during the study period.
Time Frame: 5 months: 2 months in the baseline period, one month to prep the intervention, then 2 months in the intervention period
Population: All short stay participants who had admission and discharge swabs collected and who were not co-colonized with MRSA and MSSA on admission swabs.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 101 | 120
Participants | 17 | 8

2. Secondary Outcome: Rates of Staphylococcus Aureus Transmission: Percentage of Short Stay Participants Who Acquired MRSA or MSSA (or Both) From MRSA/MSSA Transmission From Another Study Participant During the Study Period
Description: Rates of Staphylococcus aureus transmission in the baseline and intervention periods: Participants were swabbed in the anterior nares and inguinal fold at nursing home admission (or start of study period) and again at discharge (or end of study period). The DNA sequences of each SA isolate from each acquisition were evaluated to see if there was a match to another epidemiologically linked (same floor, same study period) SA isolate. This is the percentage of participants who acquired MRSA or MSSA (or both) from MRSA/MSSA transmission from another study participant during the study period.
Time Frame: 5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Intervention Period
Number analyzed (Participants) | 101 | 120
Participants | 6 | 1

ADVERSE EVENTS:
Time Frame: During the baseline period (2 months) and the intervention period (2 months)
Description: The only adverse events that were collected during the study were deaths and hospitalizations. Adverse events were assessed without regard to the specific adverse event term.
Arm/Group | Baseline Period | Intervention Period
All-Cause Mortality (participants affected / at risk) | 3/158 | 0/167
Serious Adverse Events (participants affected / at risk) | 28/158 | 28/167
Other Adverse Events (participants affected / at risk) | 0/158 | 0/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline Period (N=158) | Intervention Period (N=167)
Hospitalization (Cardiac disorders) | 1 | 3
Hospitalization (Gastrointestinal disorders) | 1 | 3
Hospitalization (General disorders) | 10 | 8
Death (General disorders) | 3 | 0
Hospitalization (Infections and infestations) | 3 | 3
Hospitalization (Nervous system disorders) | 0 | 1
Hospitalization (Psychiatric disorders) | 2 | 0
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Hospitalization (Surgical and medical procedures) | 1 | 1
Hospitalization (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT03319368/Prot_SAP_000.pdf